CLINICAL TRIAL: NCT01970150
Title: To Investigate the Effect of Application of Repeated Trans-cranial Magnetic Stimulation (rTMS) Applied on the Left Prefrontal Cortex on Electroencephalography Signal Recorded From Brain Regions Involved in Cognitive Function in Patients With Alzheimer's Disease (AD)
Brief Title: The Effect of Repeated Transcranial Magnetic Stimulation on Off-line Resting Electroencephalographic Signal in Alzheimer's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1. New data from a published trial requires substantial change in study protocol
  2. no funding available to carry the study further
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Amer Burhan, Psychiatrist, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 104382
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Alzheimer Disease
Keywords: rTMS; Alzheimer Disease; Memory; attention; EEG
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): In this intervention patients receive 5 days a week for 4 weeks of rTMS treatment with real coil
  Interventions: Device: rTMS real

INTERVENTIONS:
Device: rTMS real
  Other Names: Magstim Super Rapid 2

SUMMARY:
The purpose of this study is to examine whether the rTMS (repetitive Transcranial Magnetic Stimulation) could change cortical excitability measured by off-line EEG in Alzheimer's Disease (AD) patients.

DETAILED DESCRIPTION:
Upon meeting the inclusion criteria and providing informed consent, each participant will complete a series of 21 sessions of rTMS over the course of four weeks.During the first visit, they will be asked to undergo 1 hour of EEG (Electroencephalograph) before they start the repetitive transcranial magnetic stimulation sessions (rTMS), 0.5-hour of memory testing using MoCA and Trail Making Test (Trial A and B), 1 hour of rTMS and 1 hour of EEG after rTMS. The second visit will start approximately 24-72 hours after the first visit. During visit 2 to visit 20, participants will receive about 1 hour of TMS session 5 days a week for 4 weeks. During the 21st visit, which will be approximately one day after the last TMS session, participants will be asked to repeat 1 hour of EEG before TMS; 0.5-hour of memory testing using MoCA and Trail Making Test (Trial A and B), 1 hour TMS and 1 hour of EEG after TMS. For this study, a questionnaire concerning any potential side effects will be administrated before and after each session.

ELIGIBILITY:
Inclusion Criteria:

* Males and females,
* Age 55-85 years old,
* Able to consent and agrees to participate (if patient does not have capacity to give a consent then a caregiver will be asked )
* Fluent in English
* Diagnosed with probable AD (NINCDS-ADRDA criteria) mild stage as defined by a composite score of 1 or less on clinical dementia rating scale (CDR)

Exclusion Criteria:

* Other neurological illness that would interfere with cognitive function (significant stroke, seizure d/o, Parkinson, Huntington etc.).
* Psychiatric illness known to affect cognition such as schizophrenia/schizo-affective disorder, substance use disorder within 1 year of study, active depression or anxiety disorder or history of recurrent major mood disorder prior to cognitive change.
* Medications: benzodiazepines will be exclusionary. Other psychotropic medications including Acetyl Choline Esterase inhibitors will be allowed but the dose needs to be stable for at least one month prior to the start and during the study. Patients taking medications that might increase the risk of seizures should not participate in the study.
* Subjects with metal anywhere in the head, excluding the mouth, is generally a contraindication to TMS. This includes shrapnel, and screws and clips from surgical procedures unless the physical properties of the metal object are known and there is a strong reason for using TMS.
* Subjects with cardiac pacemakers and implanted medication pumps should not participate in most TMS studies.
* TMS also should not be performed in patients with electrodes inside the heart which might provide a low-resistance current path to electrically sensitive tissue.
* Persons with serious heart disease are at increased risk in the event of a seizure,
* Persons with increased intracranial pressure, as in acute large infarctions or trauma, are also at increased risk in the event of a seizure, and should not receive TMS.
* Pregnant women or women in child bearing age that might be pregnant.
* Patients who are already enrolled in another study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
A change in the quantitative EEG spectra in the frontal lobe, i.e. a change in percentage of theta waves, alpha and beta waves | 4 weeks
  We anticipate that rTMS exposure will result in a change in cortical excitability as evident by lowering the percentage of low frequency waves (delta and theta waves)in the cortical area under the stimulation site (left prefrontal cortex) and in functionally connected areas (contralateral cortex, inferior parietal cortex)as assessed by the EEG waves after 4 weeks of rTMS treatment.

SECONDARY OUTCOMES:
Improvement on memory and attention | 4 weeks
  We will explore the potential for improvement in memory and/or attention as asessed by MoCA and the Trail Making Test Part A and the Trail Making Test Part B, after 4 weeks of rTMS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Amer Burhan, MD, Principal Investigator — Western University, Canada
Locations (1):
- Regional Mental Health Care London, London, Ontario, Canada

REFERENCES:
- [Background] Cotelli M, Manenti R, Cappa SF, Geroldi C, Zanetti O, Rossini PM, Miniussi C. Effect of transcranial magnetic stimulation on action naming in patients with Alzheimer disease. Arch Neurol. 2006 Nov;63(11):1602-4. doi: 10.1001/archneur.63.11.1602. PMID 17101829
- [Background] Cotelli M, Manenti R, Cappa SF, Zanetti O, Miniussi C. Transcranial magnetic stimulation improves naming in Alzheimer disease patients at different stages of cognitive decline. Eur J Neurol. 2008 Dec;15(12):1286-92. doi: 10.1111/j.1468-1331.2008.02202.x. PMID 19049544
- [Background] Gawel M, Zalewska E, Szmidt-Salkowska E, Kowalski J. The value of quantitative EEG in differential diagnosis of Alzheimer's disease and subcortical vascular dementia. J Neurol Sci. 2009 Aug 15;283(1-2):127-33. doi: 10.1016/j.jns.2009.02.332. Epub 2009 Mar 6. PMID 19268969
- [Background] Schreiter Gasser U, Rousson V, Hentschel F, Sattel H, Gasser T. Alzheimer disease versus mixed dementias: an EEG perspective. Clin Neurophysiol. 2008 Oct;119(10):2255-9. doi: 10.1016/j.clinph.2008.07.216. Epub 2008 Sep 2. PMID 18768349